CLINICAL TRIAL: NCT03214328
Title: Causes of Fetal Death: Comparison of Diagnostic Accuracy Between Extensive and Selective Protocol Testing
Acronym: EMIBICI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/209/HP
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Intrauterine Fetal Death
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Determination of causes of fetal death: Both the extensive and selective protocols will be applied to each case of IUFD recruited, so that each case will serve as its own control. For each case, determination of cause from either protocol will be performed in a blind manner with respect to the other protocol.
  Interventions: Diagnostic Test: Determination of causes of fetal death

INTERVENTIONS:
Diagnostic Test: Determination of causes of fetal death — Determination of causes of fetal death using systematic protocol testing

SUMMARY:
Intrauterine fetal death (IUFD) is defined as the occurrence of fetal death at >20 weeks' gestation. IUFD affects about 1 in 160 pregnancies (6-7 per 1000 births). Optimal diagnostic evaluation for cases of IUFD is generally based on extensive protocol testing i.e. maternal and fetal blood tests, fetal bacteriology, cytogenetic analysis, autopsy, and placental examination. This extensive protocol testing may vary in clinical practice and interpretation of the results is rarely performed by multidisciplinary staff to establish cause of death. These findings are related to the fact that there are very few epidemiological studies to validate optimal protocol, no French recommendations on this subject, and a relative lack of pathologists with expertise in perinatal pathology. Only, one recent prospective study from the Netherlands has concluded that extensive protocol testing should be redefined and some diagnostics tests may only be performed with suggestive clinical circumstances. However these recommendations may not be applicable to all populations and countries. To date, there are no French published series on IUFD to evaluate causes of death in France and thereafter to better define optimal diagnostic evaluation tests. Improvement in prenatal diagnosis in France may contribute to detection of the vast majority of severe chromosomal abnormalities and malformed fetuses and particularly those at risk of death. Retrospective cohort unpublished data on IUFD from Lille and Caen have reported exceptional deaths attributable to chromosomal or malformation abnormalities. In fact in these two series, most deaths were related to placental diseases or fetal growth retardation. The hypothesis is that extensive protocol testing is not helpful in clinical practice and selective protocol testing focused on specific risk situations can be as efficient.

ELIGIBILITY:
Inclusion Criteria:

* Singleton fetus
* Intrauterine fetal death diagnosed antepartum
* Gestational age > 22 weeks
* Woman informed
* No women aged under 18 years

Exclusion Criteria:

* Pregnancy termination
* Intrapartum death
* Person placed under judicial protection, guardianship

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women underwent MFIU
Study Population: women underwent MFIU
Sampling Method: Probability Sample
Enrollment: 602 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Concordance of the causes of fetal death between selective and systematic protocol testing | an average of 6 months from fetal death

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERSPYCK, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No